CLINICAL TRIAL: NCT06075225
Title: The MAGIC Algorithm Probability Guided Preemption of Steroid-refractory Graft-versus-host Disease With Ruxolitinib
Brief Title: MAP-guided Preemptive Therapy of aGvHD by Ruxolitinib
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principle Investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HXMAP 2.0
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: GVHD; Acute Stem Cell Transplant Complications
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib is asministrated with the dose of 5mg bid for 28 days. If no signs of aGvHD, the dose of ruxolitinib is gradually tapered within the following 16 days.
  Interventions: Drug: Ruxolitinib
- Control (No Intervention): Patients assigned to the control group are treated based on symptom-triggered aGvHD therapy.

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is asministrated with the dose of 5mg bid for 28 days. If no signs of aGvHD, the dose of ruxolitinib is gradually tapered within the following 16 days.
  Arms: Ruxolitinib

SUMMARY:
The goal of this observation study is to test in patients undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT). The main question it aims to answer is:

• Effect of MAGIC algorithm probability guided preemption of aGVHD with ruxolitinib on prevention of severe aGVHD.

Participants will take ruxolitinib with the dose of 5mg bid for 28 days. If no signs of aGvHD, the dose of ruxolitinib is gradually tapered within the following 16 days.

Researchers will compare patients who don't receive preemption of aGVHD with ruxolitinib to see if there is an improvement in severe aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* Any donor type (e.g., related, unrelated, haplo) or stem cell source (bone marrow, peripheral blood, cord blood).
* Any conditioning regimen (non-myeloablative, myeloablative, or reduced intensity) is acceptable.
* GVHD prophylaxis must include a calcineurin inhibitor combined with post transplant cyclophosphamide.
* The use of serotherapy to prevent GVHD (e.g., antithymocyte globulin) prior to day 3 post-HCT is permitted
* Direct bilirubin must be <2 mg/dL unless the elevation is known to be due to Gilbert syndrome within 3 days prior to enrollment.
* ALT/SGPT and AST/SGOT must be <5 x the upper limit of the normal range within 3 days prior to enrollment.
* Signed and dated written informed consent obtained from patient or legal representative.

Exclusion Criteria:

* Patients who develop acute GVHD prior to start of study drug
* Patients at very high risk for relapse post HCT as defined by very high disease risk index
* Patients participating in a clinical trial where prevention of GVHD is the primary endpoint
* Uncontrolled active infection (i.e., progressive symptoms related to infection despite treatment or persistently positive microbiological cultures despite treatment or any other evidence of severe sepsis)
* Patients who are pregnant
* Patients on dialysis within 7 days of enrollment
* Patients requiring ventilator support or oxygen supplementation exceeding 40% FiO2 within 14 days of enrollment.
* Patients receiving investigational agent within 30 days of enrollment. However, the Principal Investigator (PI) may approve prior use of an investigational agent if the agent is not expected to interfere with the safety or the efficacy of ruxolitinib

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of High Risk Patients Who Develop Grade III or IV aGvHD | Day 100 post HCT
  Number of High Risk Patients Who Develop Grade III or IV aGvHD by day 100 post HCT

SECONDARY OUTCOMES:
Number of Participants With Non-relapse Mortality (NRM) | 6 months
  Number of participants with NRM - deaths which could not be attributed to disease relapse or progression. Nonrelapse mortality defined as death without prior relapse at 6 months
Number of Participants With Chronic GVHD Requiring Systemic Steroid Treatment | 1 year and 2 years
  Number of participants with chronic GVHD requiring systemic steroid treatment. Chronic GVHD Requiring Systemic Steroid Treatment: defined as the development of symptoms of chronic GVHD according to NIH Consensus Criteria that require treatment with oral or intravenous corticosteroids at the end of 1 year and 2 years
GvHD free and relapse free survival | 1 year and 2 years
  Survival of patients without grade 3 or 4 aGvHD or disseminated cGvHD or relapse of disease at end of 1 year post HCT at the end of 1 year and 2 years
Progression-free survival | 1 year and 2 years
  Progression-free survival of this group of patients at the end of 1 year and 2 years
Overall survival | 1 year and 2 years
  Overall survival of this group of patients at the end of 1 year and 2 years
Number of Participants With Relapse | 1 year and 2 years
  Number of participants with relapse at one year and 2 years. Relapse defined as recurrence of disease that required transplant.
Number of Participants With Serious Infections | 1 year and 2 years
  Number of participants with serious infections (defined as grade 3 by the Blood and Marrow Transplant Clinical Trials Network). Serious Infection: Defined as bacterial, fungal, viral or parasitic infections that required oral or intravenous treatments such as antibiotics
cytomegalovirus (CMV) reactivation | 1 year and 2 years
  Number of participants with cytomegalovirus (CMV) reactivation at the end of 1 year and 2 years. CMV reactivation was defined as the presence of DNA copies exceeding 10^3/ml in plasma.
grade 2 or higher hemorrhagic cystitis | 1 year and 2 years
  Number of participants with grade 2 or higher hemorrhagic cystitis at the end of 1 year and 2 years, which was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
MAGIC algorithm probability (MAP) change | Day 28 post HCT
  The change in the patient's MAGIC algorithm probability (MAP) at each time

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No